CLINICAL TRIAL: NCT05376566
Title: Hydrochloric Acid Lock Therapy for Central Line-associated Bloodstream Infections in Patients With Cancer and Hematologic Diseases
Brief Title: Hydrochloric Acid Lock Therapy for Central Line-associated Bloodstream Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Mette Bondo Mønster, Principal Investigator, Department of Paediatrics and Adolescent Medicine, Copenhagen University Hospital, Denmark, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHILD@HALT
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)
Keywords: Central line; Cancer; Lock therapy; Hydrochloric acid; Bloodstream infections; Haematological diseases
MeSH Terms: conditions — Neoplasms; Sepsis | interventions — Hydrochloric Acid; Methods; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be blinded using masked vial containing either hydrochloric acid or normal saline and coloured syringes. All masked vials have a unique three-figure randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Hydrochloric acid (2 M)
  Interventions: Drug: Hydrochloric Acid (2 M)
- Control group (Placebo Comparator): Normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hydrochloric Acid (2 M) — Hydrochloric acid (2 M) in a volume corresponding to dead space (0.3-1.8 ml) will be instilled and aspirated 10 min later; the instillation is completed 3 times.
  Other Names: Intervention
  Arms: Intervention group
Drug: Normal saline — Normal saline in a volume corresponding to dead space (0.3-1.8 ml) will be instilled and aspirated 10 min later; the instillation is completed 3 times.
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Aim: This study will test whether treatment of central line-associated bloodstream infections (CLABSI) with hydrochloric acid lock therapy (HALT) can significantly reduce the risk of treatment failure (comprising failure to clear initial infection, relapse of infection, or reinfection) in patients treated for cancer or hematologic diseases.

Study design: A multicentre, double-blinded, randomized controlled trial. Patient population: Patients (0-100 y) with cancer or a hematologic disorder and a CLABSI treated at Copenhagen University Hospital, Aarhus University Hospital, or Odense University Hospital, Denmark.

Randomization: Patients are equally assigned (1:1) to receive either HALT or placebo (normal saline). In addition to the study intervention, patients in both arms will receive standard systemic antibiotic therapy.

Sample size: A target population of 250 patients

DETAILED DESCRIPTION:
BACKGROUND

Patients with cancer or hematologic diseases and a long-term central venous access device (CVAD), including central venous catheters and intravenous ports, are at risk of developing central line-associated bloodstream infections (CLABSI). A patient with CLABSI is treated with systemic antibiotic therapy. Additionally, prompt removal of the CVAD because of CLABSI is often recommended. However, removal and replacement of a long-term CVAD is an invasive procedure and not always possible. Therefore, various types of lock therapies have been tried in attempt to cleanse and preserve the CVAD.

At more hospitals in Denmark, hydrochloric acid lock therapy (HALT) has been used routinely for patients with cancer and hematologic diseases and a CLABSI. However, HALT is not recommended outside Denmark due to limited evidence of its use.

PATIENT AND METHODS

Eligible patients with CLABSI will be enrolled during antibiotic therapy and a maximum of 5 days after the detection of a positive blood culture/CLABSI. The patients will be randomized to receive blinded lock therapy with hydrochloric acid (2 M) or placebo (normal saline). HALT and placebo lock therapy is carried out by trained oncologic nurses in identical fashion: Hydrochloric acid or normal saline in a volume corresponding to dead space (0.3-1.8ml) will be instilled and aspirated 10 min later; the instillation is completed 3 times. In addition to the study intervention, patients in both arms will receive standard systemic antibiotic therapy.

The patient is followed 6 weeks from instillation with HALT/placebo. The patient can be re-included if the patient has 1) replacement of the CVAD, or 2) a new CLABSI later than 6 weeks from a previous CLABSI. In case of re-inclusion the patient, the patient will be randomized again.

SAMPLE SIZE CALCULATION

The primary objective is to compare the risk of treatment failure between the two treatment groups.

A recent randomized, controlled trial showed a treatment failure rate of 33% within 42 days for children with CLABSI treated with placebo lock therapy (heparin in normal saline) (Wolf et al, 2018). External data from 2015-2020 of patients admitted with CLABSI and receiving HALT at Copenhagen University Hospital, Denmark, led to an estimated treatment failure rate of 17% (unpublished data).

Based on the above-estimated treatment failure rate in each group as well as feasibility constraints (incl. timeline and accrual rate), a sample size of 125 patients in each group was chosen. This choice was estimated to provide approximately 80% power to show a difference in risk between the two groups. This power was computed for a two-sided test at the type-I error level 5%, assuming a 2% dropout rate, using standard asymptotic normal approximations.

CHANGES IN THE PROTOCOL SINCE THE FIRST EDITION OF THE PROTOCOL

The first version of this protocol was published in June 2022. In October 2023, after inclusion of 61 episodes of CLABSI in paediatric patients the investigators made the following changes:

1. The titles: The word 'children' has been omitted and replaced with 'patients with cancer and hematologic diseases'.
2. Sample size: Increased from 100 to 250 patients.
3. Patient population: Changed from age 0-17 years to age 0-100 years and the inclusion of non-malignant hematologic diseases.
4. Re-inclusion of patients: Changed from 'cross-over' to new blinded randomization.
5. Time to enrolment: Changed from 48 hours to 5 days after detection of CLABSI.
6. Definition of persistent infection: Changed from "persistent positive blood cultures for more than 48 hours" to "persistent positive blood cultures 24 hours after HALT/placebo".

Reasons for changes

1. The titles:

   The titles now reflect inclusion of adults and patients with of non-malignant hematologic diseases.
2. Sample size:

   In the first power calculation, the investigators estimated a treatment failure rate in patients receiving HALT to 10%. This estimation was based on two older Danish articles, including patients in 1999-2005 (Larsen et al, 2011, Madsen et al, 2013), and data from 2010-2015 of children with CLABSI receiving HALT in Denmark (unpublished data). Recently, external data from 2015-2020 suggested a higher treatment failure rate of 17% following HALT (unpublished data). An updated power calculation using a treatment failure of 17% following HALT versus 33% following placebo suggested to increase the sample size to 250 (i.e. 125 in each group, see above).
3. The patient population:

   To meet the new sample size requirement and also address the research question in adults, the investigators will include adults from the Department of Haematology, Copenhagen University Hospital, Denmark, from October 17th, 2023. This choice was thought reasonable because: 1) External data suggest that the risk of bacteraemia in adults, and its recurrence, is similar to that observed in the paediatric population (unpublished data). 2) It is logistically feasible, as the placement and supervision of the CVADs is handled by the same anaesthesia personnel. A subgroup analysis of paediatric and adult patients will be made to complement the main analysis that will now include both paediatric and adult patients.
4. Changing of cross over in case of re-inclusion:

   In the first version of the protocol from June 2022, re-inclusion of patients was performed with cross-over design. The decision of cross-over design was mainly motivated by power considerations; it was expected to increase the power of the study. However, after re-inclusion of 10 episodes of CLABSI, the investigators realized that it led to logistical challenges and ethical issues, as it required some unblinding for the re-inclusions. The investigators have therefore changed the setup to a new randomization. The impact of this decision on the power was estimated to be very minor and therefore it was thought that such power considerations could not outweigh the importance of blinding.
5. Time to enrolment:

   The investigators have expanded the time window for including patients in the study from 48 hours after the detection of a positive blood culture to 5 days. This is because 1) new external data has shown that the risk of relapse during the first 5 days, when the patients receive antibiotic therapy, is only approximately 1% (unpublished data), 2) The expected effect of HALT is to reduce the occurrence of relapse of infection or new infection after the cessation of antibiotic treatment and 3) there is a risk of exclusion of otherwise eligible patients with a time-limit of 48 hours due to practical circumstances, e.g., during weekends.
6. Definition of persistent infection:

Definition of persistent infection is changed from "persistent positive blood cultures for more than 48 hours" to "persistent positive blood cultures 24 hours after HALT/placebo" since the installation of HALT/placebo is not always carried out immediately after the detection of a positive blood culture.

ELIGIBILITY:
Inclusion criteria

* Patients aged 0-17 years treated at pediatric oncologic department at Copenhagen University Hospital, Odense University Hospital, and Aarhus University Hospital, Denmark. Inclusion of children and adolescents from 1st of June 2022.
* Patients aged 18-100 years treated at Department of Hematology, Copenhagen University Hospital, Denmark. Inclusion of adult patients from 17th of October 2023.
* Patients receiving treatment for cancer or a hematologic disease (any type and at any point in the course of the disease).
* CVAD in situ (intravenous ports and all central lines).
* New diagnosis of CLABSI (defined as a laboratory-confirmed bloodstream infection, not secondary to infection at another site, in a patient who has a CVAD). NB, patients who had a CLABSI prior to the beginning of the study are accepted for enrollment if they have a new CLABSI during the patient enrollment phase.

The patient is followed 6 weeks from instillation with HALT/placebo. The patient can be re-included if the patient has 1) replacement of the CVAD, or 2) a new CLABSI later than 6 weeks from a previous CLABSI. In case of re-inclusion the patient, the patient will be randomized again.

Exclusion Criteria:

* Plan to remove CVAD within 6 days.
* Instantly admission to Intensive Care Uni

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Treatment failure. | Within 6 weeks after HALT or placebo (normal saline) treatment of the CVAD.
  Defined as 1) persistent infection (persistent positive blood cultures 24 hours after HALT/placebo) or relapse (a new CLABSI with an identical bacterial isolate), 2) a new CLABSI with any bacterial isolate, 3) infection-related removal of central access device (CVAD), 4) infection-related death.
  The treatment group comparison will be based on a test of the risk ratio between the two groups.

OTHER OUTCOMES:
Safety outcome 1: Infusion-related reactions i.e. anaphylactic shock, pain, rash or sensory disturbances. | Within 24 hours after start of HALT or placebo (normal saline) treatment of the CVAD.
  Incidence will be tabulated as number of events and number of patients experiencing an event according to current actual treatment.
Safety outcome 2: Death or admission to Intensive Care Unit associated to infection | Within 6 weeks after HALT or placebo (normal saline) treatment of the CVAD.
  Incidence will be tabulated as number of events, number of patients experiencing the event, and number of events per person-year of observation. Data will be categorized according to current actual treatment.
Safety outcome 3: Mechanical catheter damage or catheter occlusion requiring thrombolytic therapy. | Within 6 weeks after HALT or placebo (normal saline) treatment of the CVAD.
  Incidence will be tabulated as number of events and number of patients experiencing an event according to current actual treatment.
Exploratory outcome 1: Number of days with antibiotic treatment. | [Time Frame: Within 6 weeks after HALT or placebo (normal saline)]
  Number of days the patient was prescribed antibiotic treatment within 6 weeks after admission with CLABSI.
Exploratory outcome 2: Treatment failure | Time Frame: Within 6 weeks after HALT or placebo (normal saline)
  Defined as 1) persistent infection (persistent positive blood cultures 24 hours after HALT/placebo) or relapse (a new CLABSI with an identical bacterial isolate), 2) a new CLABSI with any bacterial isolate, 3) infection-related removal of central access device (CVAD), 4) infection-related death, 5) antibiotic treatment due to suspicion of infection despite lack of positive blood culture
  The treatment group comparison will be based on a test of the risk ratio between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrikka Nygaard, MD, ph.d., Study Chair — Department of Paediatrics and Adolescent Medicine, Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Department of Paediatrics and Adolescent Medicine, Aarhus University Hospital, Aarhus
  - Department of Haematology, Copenhagen University Hospital, Copenhagen
  - Department of Paediatrics and Adolescent Medicine, Copenhagen University Hospital, Copenhagen
  - Department of Paediatrics and Adolescent Medicine, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf J, Connell TG, Allison KJ, Tang L, Richardson J, Branum K, Borello E, Rubnitz JE, Gaur AH, Hakim H, Su Y, Federico SM, Mechinaud F, Hayden RT, Monagle P, Worth LJ, Curtis N, Flynn PM. Treatment and secondary prophylaxis with ethanol lock therapy for central line-associated bloodstream infection in paediatric cancer: a randomised, double-blind, controlled trial. Lancet Infect Dis. 2018 Aug;18(8):854-863. doi: 10.1016/S1473-3099(18)30224-X. Epub 2018 Jun 5. PMID 29884572
- [Background] Larsen LN, Malchau E, Kristensen B, Schroeder H. Hydrochloric acid treatment of tunneled central venous catheter infections in children with cancer. J Pediatr Hematol Oncol. 2011 Mar;33(2):e64-8. doi: 10.1097/MPH.0b013e3181f6933d. PMID 21285898
- [Background] Madsen M, Rosthoj S. Impact of hydrochloric acid instillation on salvage of infected central venous catheters in children with acute lymphoblastic leukaemia. Scand J Infect Dis. 2013 Jan;45(1):38-44. doi: 10.3109/00365548.2012.708941. Epub 2012 Sep 19. PMID 22992112